CLINICAL TRIAL: NCT06307483
Title: Dose-effect Relationship of Tai Chi on Health Promotion in Different Age Groups
Status: Completed | Type: Observational
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240108
Record Dates: First submitted 2024-01-24; First posted 2024-03-12 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sleep Disorder; Cardiovascular Diseases; Hypertension; Cognitive Impairment; Metabolic Disease
MeSH Terms: conditions — Sleep Wake Disorders; Cardiovascular Diseases; Hypertension; Cognitive Dysfunction; Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Taichi group: Participants in the Tai chi group were regular Tai chi practitioners who had practiced Tai chi for at least 3 months, at least three times a week for at least 30 minutes each time.
  Interventions: Behavioral: Taichi group
- Exercise group: The subjects in the exercise group had regular exercise habits, and insisted on non-Tai chi exercise for at least 3 months, at least three times a week, at least 30 minutes each time.
  Interventions: Behavioral: Exercise group
- Control group: The subjects in the control group were people without long-term exercise habits.

INTERVENTIONS:
Behavioral: Taichi group — Participants in the Tai chi group were regular Tai chi practitioners who had practiced Tai chi for at least 3 months, at least three times a week for at least 30 minutes each time.
  Groups: Taichi group
Behavioral: Exercise group — The subjects in the exercise group had regular exercise habits, and insisted on non-Tai chi exercise for at least 3 months, at least three times a week, at least 30 minutes each time.
  Groups: Exercise group

SUMMARY:
The purpose of this study is to investigate the physical and mental health status of middle-aged and elderly people of different ages and practicing Tai chi for different periods of time, so as to provide a strong theoretical basis and practical guidance for delaying age-related aging and preventing and treating the occurrence and development of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20-79 years.
* People who practice Tai chi for a long time.
* People with long-term exercise habits.
* People who have no habit of exercising.

Exclusion Criteria:

* People currently participating in other interventions (e.g., nutrition, psychological, exercise, health education).
* People with cognitive impairment and movement disorders.
* Cardiovascular and cerebrovascular events (physician-diagnosed heart disease, such as coronary heart disease, hypertensive heart disease, acute myocarditis, pulmonary heart disease, etc.) in the past 6 months.
* People with other serious chronic diseases, such as asthma, cancer, chronic heart failure, severe depression, or other mental disorders.

Ages: 20 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects were people of both sexes aged 20-79 years with long-term Tai chi practice habit or long-term exercise habit or no exercise habit.
Sampling Method: Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  With subscale scores ranging from 0 to 3, the PSQI assesses subjective sleep quality in the previous month and consists of seven items (sleep duration, sleep latency, sleeping medications, sleep disturbance, daytime dysfunction, sleep quality, and sleep efficiency). The total score of the PSQI, ranging from 0 to 21, is the sum of subscale scores, and the higher the scores, the lower the subjective quality of sleep.
Heart rate variability (HRV) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  HRV, a non-invasive method used to evaluate the autonomic nervous system modulation on the cardiac sinus node, describes the oscillations between consecutive electrocardiogram R-R intervals. High levels of HRV indices are generally signs of efficient autonomic mechanisms that characterise a healthy individual, while low or reduced HRV often show an autonomic nervous system malfunction and may imply health impairment.
Flow-mediated dilation (FMD) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Flow-mediated dilation (FMD) can assess endothelium-dependent vasodilation, evaluating vascular elasticity and dilation function. Its mechanism involves inducing reactive hyperemia, increasing arterial blood flow, leading to elevated shear stress on the vessel wall, prompting endothelial cells to release NO, resulting in vasodilation. A normal FMD value is ≥7%; values <4% indicate endothelial dysfunction.
Cardiac Output (CO) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Cardiac Output (CO) is a key indicator in echocardiographic examinations, used to measure the total volume of blood pumped by the heart per minute. This parameter reflects the efficiency of the heart's pumping action and the status of systemic blood circulation. The measurement of Cardiac Output is based on the volume of blood ejected by the heart with each beat (stroke volume) and the number of heartbeats per minute. Cardiac Output is typically expressed in liters per minute (L/min).
Intima-Media Thickness (IMT) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Intima-Media Thickness (IMT) is a significant indicator measured through carotid ultrasound examination, used to assess the thickness of the carotid artery wall. The measurement of IMT focuses on the distance between the intima and media layers of the carotid artery, serving as a key indicator of early changes in atherosclerosis.
The Berg Balance Scale（BBS） | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The BBS scale evaluates an individual's ability to maintain their balance while performing functional activities. It includes 14 items and each section is scored between 0 (worst) and 4 (best), and measures level of dependence/independence in positions such as standing from sitting, standing with feet together, standing in full balance position, balancing on one leg, as well as ability to change positions. High BBS score indicates good balance. Participants are classifed based on BBS score as high fall risk, balance disorder (0-20 points), moderate fall risk, acceptable balance (21-40 points), and low fall risk, good balance (41-56 points)
The 30-s Chair Stand Test | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  In the 30-s CST, which assesses dynamic balance and physical ftness, the individual sits in the middle of a chair with seat height of 43 cm, with a straight back, feet fat on the foor, and arms crossed over the chest with hands at shoulder level. The test starts with the subject in this position at the "go" command. The number of times the patient rises to a full standing position without assistance in 30 s is recorded as the test score. A score of 5 indicates strength and 10 indicates both strength and endurance
Lower limb muscle strength test | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Using the micro FET3 (HOGGAN, USA) to test lower limb muscle strength. The main muscles tested include the tibialis anterior, triceps surae, quadriceps femoris, hamstrings, and iliopsoas. Each muscle is tested twice, and the maximum value is recorded

SECONDARY OUTCOMES:
Body Fat Percentage | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Body fat percentage refers to the proportion of body fat weight in the total body weight of the human body, which reflects the amount of fat content in the human body. Normal adult body fat percentage should be kept in a certain range. A high body fat percentage can be considered a criterion for obesity.
Finger-Ring Test | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The finger-ring test is an effective alternative to calf circumference, in which people encircle the thickest part of the non-dominant calf with the index fingers and thumbs of both hands, and are at an increased risk of developing sarcopenia if the measured calf fits just right or is turned smaller than their fingers.
Hand Grip Strength | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Grip strength is mainly a test of the degree of development of the upper limb muscle groups, testing the subject's forearm and hand muscle strength, reflecting the level of development of the human body's upper limb strength of an indicator.
Upper and Lower Body Flexibility | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Flexibility is often considered one of the most important components of physical fitness. It is often used to describe the range of motion of a single joint or a series of joints. Among the most commonly reported simple field tests of flexibility of the lower extremity have been sit and reach (SR) test.
The SARC-F scale | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The SARC-F scale is a screening tool for muscle wasting disorders that has been developed in recent years to provide a rapid assessment of muscle strength and function without the need to rely on expensive instrumentation to measure muscle mass. SARC-F ≥ 4 is defined as sarcopenia. The questions of SARC-F cover physical functions targeting sarcopenia or initial presentation for sarcopenia.
Shape Trail Test (STT) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The Trail Making Test (TMT) scoring is expressed in terms of the time in seconds for Part A and Part B of the test. Some examiners also calculate a Trails B/Trails A ratio. The TMT is one of the most sensitive and popular tests for identifying mild cognitive impairment and mild dementia. It measures the speed for attention, sequencing, mental flexibility, and of visual search and motor function, mainly reflecting the ability of "set shifting".In China, the Shape Trail Test (STT) is more widely used. The STT was developed with the intent to minimize cultural bias and provide a more accurate cognitive measure in diverse populations.In the STT,Part B shows all numbers (from 1 to 25) twice, once in a circle and once in a square. The participants are asked to make lines alternating between circles and squares and disregarding the numbers of the alternate shapes.
  The scoring of the STT has several indexes: (1) time in seconds required to complete each par
1-back Task more-odd shifting Task Stroop Task | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The 1-back task was used to explore the performance of different age groups on the memory updating task. subjects were used to investigate the relationship between physical activity and the executive function in the elderly by using the International Physical Activity Scale, 1-back Task, more-odd shifting Task and Stroop Task. E-Peime3.0 software was used to present the above paradigm, and SPSS20.0 software was used to analyze the response time and accuracy of the subjects.
Timed Up and Go | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The Timed up and go test (TUGT) was used to assess functional mobility. Participants were asked to walk at their ordinary walking speed during the tes t. They were seated at the beginning of the test and were asked to stand up from the chair, walk 3 m, turn around, return to the chair, and sit down again. The duration between rising from the chair and sitting down was measured with a stopwatch
Close-eyed stepping in place | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Prepare to draw a 20 cm x 20 cm square on the ground with chalk. The subject is required to stand in the center of the square and, upon hearing a command, perform stepping in place with eyes closed. The timing stops if the subject steps on the line or exits the square while stepping with eyes closed. The test should be conducted twice, and the longest time taken should be recorded
Single-leg stance with eyes closed | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  For this test, the subject wears comfortable flat shoes, places hands on hips, and closes their eyes. They then stand on each leg separately, with the other leg bent at the knee and lifted 10cm off the ground, with the lower leg touching the standing leg (although it can be slightly apart during the test). Timing begins when the foot leaves the ground and ends if the standing foot moves, the body leans significantly, or the lifted foot touches the ground. The test is conducted 3 times, with a 1-minute rest in between, and the best result is recorded
Ankle-Brachial Index (ABI) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Ankle-Brachial Index (ABI) is a non-invasive vascular test that assesses peripheral arterial disease by comparing blood pressure measurements in the ankles and arms. ABI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm. A normal ABI value is typically between 0.90 and 1.30, with lower values indicating potential arterial blockages. ABI is a crucial diagnostic tool for evaluating peripheral arterial health and identifying risks associated with reduced blood flow to the extremities.
Short-Physical Performance Battery (SPPB) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The SPPB is the National Institute on Aging's approved method of assessing muscle function in older adults. There are three components, the balance test, the gait speed test, and the chair sit-to-stand test. Asian Working Group for Sarcopenia: 2019 Consensus (AWGS) 2019 recommends SPPB score ≤9 as the cutoff for low physical performance.
Hospital Anxiety and Depression Scale (HADS) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The Hospital Anxiety and Depression Scale (HADS) was devised 30 years ago by Zigmond and Snaith to measure anxiety and depression in a general medical population of patients. In this study, it was used to measure the mental condition of participants. The scale comprises 14 questions which related 2 underlying sub-scale dimensions, anxiety (HADS-A) and depression (HADS-D) respectively. Each subscale has 7 items and each item is scored with 0-3 points. The minimum and maximum values of the HADS are 0 and 42. The higher the score, the more severe the condition is. The minimum and maximum values of the subscales are 0 and 21, and higher scores mean a worse outcome. Those with score ≥8 on HADS-A or HADS-D were considered to be at high risk of having anxiety or depression.
Blood pressure variability (BPV) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  BPV is defined as a change in the value of arterial blood pressure over a defined period of time. Multiple studies have shown that BPV is a strong and independent risk factor for cardiovascular diseases (CVDs), chronic kidney disease, dementia, and stroke, as well as hypertension-related morbidity and mortality.
HUR Labs Balance Software Suite | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Use the HUR Labs Balance Software Suite static balance testing system to conduct static balance capacity testing. The testing protocol includes Romberg30s, single-leg stance with eyes closed, and Limits of Stability (LOS) testing with a star balance test
E/A ratio | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  The E/A ratio is an important indicator in echocardiography used to assess blood flow between the left atrium and the left ventricle of the heart. It is calculated using two-dimensional Doppler ultrasound technology by measuring the velocity of blood flow during the early phase of ventricular relaxation (E wave) and during atrial contraction (A wave). The E/A ratio reflects the diastolic function of the heart, particularly the filling pressures and filling rates of the left ventricle.
Star Excursion Balance Test apparatus（SEBT） | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Using a tape measure, mark a "zero" point on the ground and measure out 8 directions at 45° intervals, and assign names to each direction. For the test, the subject should first lie on a yoga mat for the measurement of leg length. Then, the subject should stand in the center, with hands on hips, supporting leg bent at the knee, and the non-supporting leg should be extended as far as possible in 5 directions on the same side. The test should be conducted twice, and the best score should be used. There are two standardized calculation methods: one method calculates the total score as (the sum of the maximum values in the 8 directions) / (8 times the leg length) × 100; the other method calculates the relative distance in each direction as the maximum distance reached / leg length × 100
Montreal Cognitive Assessment(MoCA) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  the Montreal Cognitive Assessment(MoCA) was specifically developed as a screening tool for MCI and mild dementia, and has been shown to have high sensitivity and specificity for differentiating individuals with MCI from healthy individuals.A higher score indicates better cognitive function. Firstly, MCI was determined according to the cut point values of different educational levels.Total score ≤13 (below primary school), ≤19 (1~6 years of education), ≤24 (≥7 years of education).
Brachial-ankle pulse wave velocity (BaPWV) | This study was a cross-sectional study. Each subject was measured only once from the day of randomization to the first assessment, assessed up to 3 months
  Brachial-ankle pulse wave velocity (BaPWV) is a non-invasive measure of arterial stiffness, reflecting the speed of the arterial pressure wave between the brachial artery and ankle arteries. Higher BaPWV values indicate increased arterial stiffness, associated with cardiovascular risks such as hypertension and atherosclerosis. It serves as a valuable tool in clinical settings for assessing vascular health, predicting cardiovascular events, and monitoring the effectiveness of interventions to improve arterial elasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No